CLINICAL TRIAL: NCT01755559
Title: Efficacy of Artesunate-amodiaquine, Dihydroartemisinin-piperaquine and Artemether-lumefantrine Combination Therapies for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Children Aged 6 to 59 Months in Maradi, Niger 2012-13
Brief Title: Efficacy of Three ACTs for the Treatment of Falciparum Malaria in Maradi Niger
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Centre de Recherche Médicale et Sanitaire (Cermes), Niamey (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Epicentre/Nig/2012/Palu3ACT
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Malaria
Keywords: malaria; artemisinin; artemisinin-based combination therapies; Plasmodium falciparum; efficacy
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Artesunate-amodiaquine (Other): Efficacy estimates at 95%
  Interventions: Drug: Artesunate-amodiaquine
- Dihydroartemisinin-piperaquine (Other): Efficacy estimates at 95%
  Interventions: Drug: Dihydroartemisinin-piperaquine
- Artemether-lumefantrine (Other): Efficacy estimates at 95%
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artesunate-amodiaquine — antimalarial ACT
  Other Names: AS-AQ Winthrop® Sanofi Aventis
  Arms: Artesunate-amodiaquine
Drug: Dihydroartemisinin-piperaquine — antimalarial ACT
  Other Names: Euratesim, Sigma-Tau
  Arms: Dihydroartemisinin-piperaquine
Drug: Artemether-lumefantrine — antimalarial ACT
  Other Names: Coartem, Novartis
  Arms: Artemether-lumefantrine

SUMMARY:
Study treatments:

* Artemether-lumefantrine
* Artesunate-amodiaquine
* Dihydroartemisinin-piperaquine

Location:

Maradi, Niger

Principal Objective:

To measure the clinical and parasitological efficacy of the three artemisinin combination therapies over a period of 42 days from the start of treatment and with polymerase chain reaction assay (PCR) adjustment.

Secondary objectives:

* To determine the blood concentration of the non-artemisinin component of the treatment (lumefantrine, desethylamodiaquine or piperaquine) at day 7
* To assess the incidence of adverse events during the follow-up period;
* To measure speed of parasite clearance

Methods:

In vivo non comparative study as for WHO standardised protocol. The study also measure the concentration of the non-artemisinin component.

Target population:

Children under 5 years of age consulting the integrated health centres of Andoumé and Dix-sept portes in Maradi.

Sample size:

221 patients per study treatment; 663 patients in total.

Treatment allocation:

Random.

Outcomes:

* Early treatment failure,
* Late clinical failure,
* Late parasitological failure,
* Adequate clinical and parasitological response.

Analysis:

* Cumulative success or failure rate (Kaplan-Meier analysis).
* Proportions of early treatment failures, late clinical failures, late parasitological failures, and adequate clinical and parasitological response (called also Per-protocol analysis).

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 59 months
* Weight ≥ 5 kg
* Mono-infection with P. falciparum detected by microscopy
* Parasitic density between 2,000 and 200,000 asexual forms /µL of blood
* Axillary temperature ≥ 37.5°C or history of fever during the previous 24 hours
* Ability and willingness to comply with the protocol for the duration of the study and to comply with the study visit schedule (home is within one hour of walk from the outpatient department, no near-term travel plans, etc.)
* Consent of a parent or guardian who is at least 18 years of age.

Exclusion Criteria:

* Presence of general danger signs as defined by the WHO,
* Presence of signs of severe malaria according to the definitions of WHO,
* Severe anemia (haemoglobin <5 g/dL),
* Known history of symptomatic cardiac arrhythmias or with clinically relevant bradycardia,
* Family history of sudden death or of congenital prolongation of corrected QT interval,
* Use of antiarrhythmics or neuroleptics,
* Known history of hypersensitivity to any of the study medications,
* Severe malnutrition (defined as a weight-height ratio of < -3 z-score according to the 2006 WHO reference (20) and / or a mid-upper arm circumference lower than 115 mm and / or the presence of symmetrical oedema of the feet),
* Presence of a febrile condition due to a disease other than malaria (i.e. measles, acute lower respiratory tract infection, otitis media, tonsillitis, abscess, severe diarrhoea with dehydration, etc.)
* History of a full treatment course with one of the three study drugs in the past 28 days. The prior incomplete intake of one of the three study drugs or prior intake of antimalarial drugs not being tested in the study does not exclude a patient from participating in this study. However, information on these previous treatments will be carefully recorded.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 663 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Adequate clinical and parasitological response | 42 days after treatement start
  Absence of parasitaemia on day 42, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure.

SECONDARY OUTCOMES:
Early treatment failure | 1 to 3 days after tratment start
  * General danger signs or signs of severe malaria on days 1, 2, or 3, in the presence of parasitaemia , or
  * Parasitaemia on day 2 higher than on day 0, irrespective of axillary temperature, or
  * Parasitaemia on day 3 with axillary temperature ≥ 37.5°C, or
  * Parasitaemia on day 3 ≥ 25% count on day 0 irrespective of axillary temperature.
Late clinical failure | from day 4 to day 42 after treatment start
  * General danger signs or severe malaria in the presence of parasitaemia on any day between day 4 and day 42 in patients who did not previously meet any of the criteria of early treatment failure; or
  * Presence of parasitaemia on any day between day 4 and day 42 with axillary temperature ≥ 37.5 °C in patients who did not previously meet any of the criteria of early treatment failure.
Late Parasitological Failure | from day 7 to day 42 after treatment start
  - Presence of parasitaemia on any day between day 7 and day 42 with axillary temperature < 37.5 °C in patients who did not previously meet any of the criteria of early treatment failure or late clinical failure.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Grandesso, MSc, Principal Investigator — Epicentre; Lynda Woi Messe, MD, Study Chair — Epicentre; Ibrahim M Laminou, PhD, Study Chair — Cermes; Jean-François Etard, PhD, Study Chair — Epicentre
Locations (1):
- Andoumé Health Centre, Maradi, Maradi Region, Niger

REFERENCES:
- [Derived] Grandesso F, Guindo O, Woi Messe L, Makarimi R, Traore A, Dama S, Laminou IM, Rigal J, de Smet M, Ouwe Missi Oukem-Boyer O, Doumbo OK, Djimde A, Etard JF. Efficacy of artesunate-amodiaquine, dihydroartemisinin-piperaquine and artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria in Maradi, Niger. Malar J. 2018 Jan 25;17(1):52. doi: 10.1186/s12936-018-2200-1. PMID 29370844